CLINICAL TRIAL: NCT05133674
Title: Therapeutic Dose Monitoring (TDM) of Tamoxifen and Its Active Metabolites in Combination With Patient-reported Symptom Scores Among Patients With Breast Cancer Receiving Adjuvant Tamoxifen Treatment
Brief Title: Therapeutic Dose Monitoring (TDM) of Tamoxifen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Elham Hedayati, MD, PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDM of TAM
Record Dates: First submitted 2021-10-07; First posted 2021-11-24 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Breast Carcinoma; Breast Tumors; Cancer of Breast; Malignant Neoplasm of Breast
Keywords: Adjuvant Tamoxifen; Endoxifen; Patient reported outcomes; Adjuvant endocrine treatment; Selective Estrogen Receptor Modulators
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 0 (Experimental): Blood concentrations of tamoxifen, 4-hydroxytamoxifen and Z-endoxifen will be measured.
  Interventions: Drug: Tamoxifen 20 mg

INTERVENTIONS:
Drug: Tamoxifen 20 mg — i) a self-testing capillary kit, the rhelise™ kit for measuring the concentrations of tamoxifen, 4-hydroxytamoxifen and Z-endoxifen and ii) a patient interactive digital tool (app) mBraze to collect data about symptoms and guide breast cancer patients on adjuvant tamoxifen.

SUMMARY:
Tamoxifen is a potent and effective drug reducing the risk of dying from breast cancer in the adjuvant setting. Although more modern drugs have partly replaced tamoxifen, it is helpful in the neoadjuvant and metastatic settings as a single drug. Despite that, in the adjuvant setting, it is a valuable drug.

This study aims to validate and study the feasibility of serial assessments, including therapeutic drug monitoring of tamoxifen, 4-hydroxytamoxifen and Z-endoxifen by capillary blood sampling, combined with patient-reported symptom scores. This will provide preliminary data to allow us to develop a future multicentre randomised clinical trial of personalised dose monitoring and adjustment of adjuvant tamoxifen therapy to enhance the quality of life and breast cancer outcomes.

DETAILED DESCRIPTION:
This repeated-measures, prospective, open-label, single-centre study is designed for women with stage 0-3 breast cancer receiving adjuvant tamoxifen 20 mg/day.

Inclusion criteria:

1. Female patients aged ≥ 18 years with hormone-positive stage 0-3 breast cancer.
2. Performance status Eastern Cooperative Oncology Group (ECOG) 0-2.
3. Ongoing daily adjuvant tamoxifen minimum of 2 months ± gonadotropin-releasing hormone (GnRH) analogues ± radiation therapy (RT) for stage 3 breast cancer.
4. Locally recurrent disease, previously treated with adjuvant tamoxifen.
5. Able to use software applications developed specifically for small, wireless computing devices, such as smartphones and tablets.
6. Have small, wireless computing devices, such as smartphones and tablets.

Exclusion Criteria:

1. Fulfilling any of the contraindications for tamoxifen.
2. Metastatic (stage IV) breast cancer.
3. Included in other clinical studies receiving not approved investigational medicinal drug.
4. Ongoing pregnancy or lactation.
5. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

No. Of Subjects: 40 female subjects.

Measured components: Tamoxifen, 4-hydroxytamoxifen and Z-endoxifen

Study design: Blood samples for measurement of tamoxifen, 4-hydroxytamoxifen and Z-endoxifen will be drawn capillary in total at 4-time points, at inclusion (baseline), and after 1, 2, and 3 weeks for each participant; and venously in total at 2-time points, at inclusion (baseline), and after 3 weeks for each participant.

At each time, participants will be asked to leave 2 vials of capillary blood (50ul x2) using the rhelise™ kit and 2 samples of conventional venous blood for blood and plasma (5 ml x 2).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥ 18 years with hormone-positive stage 0-3 breast cancer.
2. Performance status ECOG 0-2.
3. Ongoing daily adjuvant tamoxifen minimum of 2 months ± GnRH analogues ± RT for stage 3 breast cancer.
4. Locally recurrent disease, previously treated with adjuvant tamoxifen.
5. Able to use software applications developed specifically for small, wireless computing devices, such as smartphones and tablets.
6. Have small, wireless computing devices, such as smartphones and tablets.

Exclusion Criteria:

1. Fulfilling any of the contraindications for tamoxifen.
2. Metastatic (stage IV) breast cancer.
3. Included in other clinical studies receiving not approved investigational medicinal drug.
4. Ongoing pregnancy or lactation.
5. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
To validate the rhelise™ kit for monitoring tamoxifen, 4-hydroxytamoxifen and Z-endoxifen among patients recommended or who have ongoing adjuvant tamoxifen. | At at inclusion (baseline) for each participant.
  Blood concentrations of tamoxifen, 4-hydroxytamoxifen and Z-endoxifen at baseline, two weeks, 1, 2, and 3 weeks by capillary and venous blood sampling (whole blood/plasma).
To validate the rhelise™ kit for monitoring tamoxifen, 4-hydroxytamoxifen and Z-endoxifen among patients recommended or who have ongoing adjuvant tamoxifen. | At week 3 after inclusion for each participant.
  Blood concentrations of tamoxifen, 4-hydroxytamoxifen and Z-endoxifen at baseline, two weeks, 1, 2, and 3 weeks by capillary and venous blood sampling (whole blood/plasma).

SECONDARY OUTCOMES:
To test the correlations of concentrations found in the capillary sample (rhelise™ kit) and the venous blood sample (gold standard). | At 4-time points, at inclusion (baseline), and after 1, 2, and 3 weeks for each participant.
  Correlations of blood concentrations of tamoxifen, 4-hydroxytamoxifen and Z-endoxifen between venous blood samples and capillary blood samples (Sensitivity and specificity).
To validate user acceptability and feasibility of self-testing the capillary kit. | At 4-time points, at inclusion (baseline), and after 1, 2, and 3 weeks for each participant.
  Capillary blood test concentrations of tamoxifen, 4-hydroxytamoxifen and Z-endoxifen were taken by the patient and the research nurse.
Symptom distresses scores measured by the patient interactive digital tool (application) mBraze. | at baseline and 3 weeks.
To compare and correlate blood concentrations of tamoxifen, 4-hydroxytamoxifen and Z-endoxifen with patient-reported outcome measures and the application mBraze for symptom self-monitoring. | at baseline and 3 weeks
  Correlations between tamoxifen, 4-hydroxytamoxifen and Z-endoxifen concentrations and symptom distress score ((fatigue, insomnia, pain, body image, and systemic therapy side-effect and cognitive-, emotional-, role-, sexual and social functioning).
  Correlations between tamoxifen, 4-hydroxytamoxifen and Z-endoxifen concentrations and symptom distress in the same patient.
To validate the user experience of the mBraze app. | at 3 weeks.
  - The interview on user acceptability and attitudes toward mBraze.
To validate the usability of the mBraze app. | at 3 weeks.
  - Self-reported usability and user experience of the mBraze app measured with system usability scale (SUS).
To determine user acceptability and attitudes toward self-testing. | at 3 weeks.
  - The interview on user acceptability and attitudes toward self-testing.

CONTACTS AND LOCATIONS:
Overall Officials: Elham Hedayati, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Davies C, Godwin J, Gray R, Clarke M, Cutter D, Darby S, McGale P, Pan HC, Taylor C, Wang YC, Dowsett M, Ingle J, Peto R. Relevance of breast cancer hormone receptors and other factors to the efficacy of adjuvant tamoxifen: patient-level meta-analysis of randomised trials. Lancet. 2011 Aug 27;378(9793):771-84. doi: 10.1016/S0140-6736(11)60993-8. Epub 2011 Jul 28. PMID 21802721
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Aromatase inhibitors versus tamoxifen in early breast cancer: patient-level meta-analysis of the randomised trials. Lancet. 2015 Oct 3;386(10001):1341-1352. doi: 10.1016/S0140-6736(15)61074-1. Epub 2015 Jul 23. PMID 26211827
- [Background] Eriksson M, Eklund M, Borgquist S, Hellgren R, Margolin S, Thoren L, Rosendahl A, Lang K, Tapia J, Backlund M, Discacciati A, Crippa A, Gabrielson M, Hammarstrom M, Wengstrom Y, Czene K, Hall P. Low-Dose Tamoxifen for Mammographic Density Reduction: A Randomized Controlled Trial. J Clin Oncol. 2021 Jun 10;39(17):1899-1908. doi: 10.1200/JCO.20.02598. Epub 2021 Mar 18. PMID 33734864
- [Background] He W, Fang F, Varnum C, Eriksson M, Hall P, Czene K. Predictors of Discontinuation of Adjuvant Hormone Therapy in Patients With Breast Cancer. J Clin Oncol. 2015 Jul 10;33(20):2262-9. doi: 10.1200/JCO.2014.59.3673. Epub 2015 Jun 1. PMID 26033800
- [Background] Madlensky L, Natarajan L, Tchu S, Pu M, Mortimer J, Flatt SW, Nikoloff DM, Hillman G, Fontecha MR, Lawrence HJ, Parker BA, Wu AH, Pierce JP. Tamoxifen metabolite concentrations, CYP2D6 genotype, and breast cancer outcomes. Clin Pharmacol Ther. 2011 May;89(5):718-25. doi: 10.1038/clpt.2011.32. Epub 2011 Mar 23. PMID 21430657
- [Background] Fabian CJ. Will a Low-Dose Option Improve Uptake of Tamoxifen for Breast Cancer Risk Reduction? J Clin Oncol. 2019 Jul 1;37(19):1595-1597. doi: 10.1200/JCO.19.00656. Epub 2019 May 13. No abstract available. PMID 31082270
- [Background] Smith SG, Sestak I, Forster A, Partridge A, Side L, Wolf MS, Horne R, Wardle J, Cuzick J. Factors affecting uptake and adherence to breast cancer chemoprevention: a systematic review and meta-analysis. Ann Oncol. 2016 Apr;27(4):575-90. doi: 10.1093/annonc/mdv590. Epub 2015 Dec 8. PMID 26646754
- [Background] Thoren L, Lindh JD, Ackehed G, Kringen MK, Hall P, Bergh J, Molden E, Margolin S, Eliasson E. Impairment of endoxifen formation in tamoxifen-treated premenopausal breast cancer patients carrying reduced-function CYP2D6 alleles. Br J Clin Pharmacol. 2021 Mar;87(3):1243-1252. doi: 10.1111/bcp.14500. Epub 2020 Aug 9. PMID 32713032
- [Background] Borges S, Desta Z, Li L, Skaar TC, Ward BA, Nguyen A, Jin Y, Storniolo AM, Nikoloff DM, Wu L, Hillman G, Hayes DF, Stearns V, Flockhart DA. Quantitative effect of CYP2D6 genotype and inhibitors on tamoxifen metabolism: implication for optimization of breast cancer treatment. Clin Pharmacol Ther. 2006 Jul;80(1):61-74. doi: 10.1016/j.clpt.2006.03.013. PMID 16815318
- [Background] Jin Y, Desta Z, Stearns V, Ward B, Ho H, Lee KH, Skaar T, Storniolo AM, Li L, Araba A, Blanchard R, Nguyen A, Ullmer L, Hayden J, Lemler S, Weinshilboum RM, Rae JM, Hayes DF, Flockhart DA. CYP2D6 genotype, antidepressant use, and tamoxifen metabolism during adjuvant breast cancer treatment. J Natl Cancer Inst. 2005 Jan 5;97(1):30-9. doi: 10.1093/jnci/dji005. PMID 15632378
- [Background] Ferraldeschi R, Newman WG. The Impact of CYP2D6 Genotyping on Tamoxifen Treatment. Pharmaceuticals (Basel). 2010 Apr 15;3(4):1122-1138. doi: 10.3390/ph3041122. PMID 27713292
- [Background] Cronin-Fenton DP, Damkier P. Tamoxifen and CYP2D6: A Controversy in Pharmacogenetics. Adv Pharmacol. 2018;83:65-91. doi: 10.1016/bs.apha.2018.03.001. Epub 2018 May 7. PMID 29801584
- [Background] Sanchez-Spitman AB, Swen JJ, Dezentje VO, Moes DJAR, Gelderblom H, Guchelaar HJ. Effect of CYP2C19 genotypes on tamoxifen metabolism and early-breast cancer relapse. Sci Rep. 2021 Jan 11;11(1):415. doi: 10.1038/s41598-020-79972-x. PMID 33432065
- [Background] Bergqvist J, Lundstrom S, Wengstrom Y. Patient interactive digital support for women with adjuvant endocrine therapy in order to increase compliance and quality of life. Support Care Cancer. 2021 Jan;29(1):491-497. doi: 10.1007/s00520-020-05476-z. Epub 2020 May 13. PMID 32405965